CLINICAL TRIAL: NCT03595956
Title: Transgender Cohort Study of Gender Affirmation and HIV-related Health
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fenway Community Health (Other)
Collaborators: Callen-Lorde Community Health Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sari Reisner, ScD, Director of Transgender Research & Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1239849
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: HIV/AIDS; STI; Gender Dysphoria; Transsexualism; Gender Identity; Depression, Anxiety
Keywords: Transgender; HIV/AIDS; Gender affirmation; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Gender Dysphoria; Transsexualism; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Gender Affirmation (MGA) Cohort: Patients engaged in gender-affirming care.
  Interventions: Other: Medical gender affirmation

INTERVENTIONS:
Other: Medical gender affirmation — The intervention to be evaluated is medical gender affirmation delivered in primary care (medical gender affirmation: hormones and/or surgery vs none).

SUMMARY:
This observational research study will evaluate medical gender affirmation delivered in primary care as an intervention to reduce disparities in HIV-related outcomes (e.g., low rates of PrEP uptake for HIV-uninfected patients, high rates of viral suppression for HIV-infected patients) for transgender patients in two urban federally-qualified community health centers.

DETAILED DESCRIPTION:
This observational, longitudinal prospective cohort study will evaluate whether medical gender affirmation delivered in primary care improves HIV-related outcomes for transgender patients. Medical gender affirmation therapies-hormones and surgical interventions-are medically necessary treatments shown to improve psychological functioning and quality of life for transgender patients. It is not yet known whether these treatments improve HIV-related outcomes over time because studies providing the best evidence of medical gender affirmation's clinical effectiveness do not examine HIV-related outcomes in transgender adult patients. To fill this gap, the proposed study will prospectively evaluate the effects of medical gender affirmation delivered in primary care on HIV-related outcomes in a multi-site clinic-based cohort of 4,500 diverse transgender patients from two urban U.S. health centers who are leaders in transgender healthcare. Transgender adult primary care patients at Fenway Health in Boston, MA and Callen-Lorde Community Health Center in New York City, NY will be enrolled over 12 months and followed prospectively for 12 months. Bio-behavioral data will be linked, including electronic patient-reported outcomes (baseline, 6-month, 12-month assessments), and electronic health record (EHR) data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Have a gender identity differing from their assigned sex at birth (verified at screening via two-step method cross-categorizing natal sex and gender identity);
* Current or new primary care patient at Fenway Health or Callen-Lorde Community Health Center (primary care patients are defined as those who had at least one medical visit in a 12-month period);
* Able to read, speak, and understand English and/or Spanish;
* Willing and able to provide informed consent.

Exclusion Criteria:

* Under 18 years of age;
* Unable to read, speak, and understand English and/or Spanish;
* Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must have a gender identity differing from their assigned sex at birth (verified at screening via two-step method cross-categorizing natal sex and gender identity).
Study Population: A total of 4,500 participants (46% people of color; 45% transgender women, 33% transgender men; 22% nonbinary individuals) will be enrolled across both study sites.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Viral suppression in HIV-infected transgender patients | 12 months
  Longitudinally evaluate whether medical gender affirmation in primary care (i.e., hormones and/or surgical interventions) improve HIV outcomes (i.e., viral suppression) in transgender adult patients over 12 months of follow-up. Medical gender affirmation is operationalized as a dichotomous variable (binary: hormones and/or surgery vs. none); viral suppression is defined as <200 copies/mL (Yes/No).
Uptake of pre-exposure prophylaxis (PrEP) in HIV-uninfected transgender patients | 12 months
  Longitudinally evaluate whether medical gender affirmation in primary care (i.e., hormones and/or surgical interventions) improve HIV prevention (i.e., PrEP uptake) in transgender adult patients over 12 months of follow-up. Medical gender affirmation is operationalized as a dichotomous variable (binary: hormones and/or surgery vs. none); PrEP uptake is a dichotomous variable (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Sari Reisner, ScD, Principal Investigator — Brigham and Women's Hospital & Harvard Medical School
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD may be available to outside individuals by contacting the principal investigator (PI). The first will be after all of the baseline data is collected. The investigators will institute a concept plan process where internal study staff first have the availability to write primary papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, the investigators may welcome this collaboration. A similar process will happen for outcome data; however this will not be possible until the publication and release of the outcome paper(s). Information regarding the availability of data for analysis will be listed on the PI's web page. Contact information for the PI will be listed in all manuscripts and publications as another means to access data.
Supporting Information: Study Protocol, ICF